CLINICAL TRIAL: NCT07259486
Title: Comparison of Outcomes of Early Kangaroo Mother Care and Standard Method Care in Healthy Low Birth Weight Preterm Neonates at a Tertiary Care Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Komal Khadim Hussain, Senior Medical Officer, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB/2022/921/SIMS
Record Dates: First submitted 2025-09-28; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: To Compare the Outcomes of Early Kangaroo Mother Care and Standard Method Care in Healthy Low Birth Weight Preterm Neonates; Premature
MeSH Terms: conditions — Premature Birth | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial study was conducted in low birth weight babies admitted in Services Hospital Lahore, Punjab, Pakistan. Inclusion criteria were neonate with birth weight 1250 to 1800 gm., gestational age >30weeks to <37 weeks and the hemodynamically stable after birth. A detailed history was taken from the mother/caregiver and from an obstetric record and then entered in the structured questionnaire. Gestational age was determined by best obstetric estimates and new Ballard score. Exclusion criteria were a major life-threatening congenital malformation, severe perinatal asphyxia, babies require a ventilator or inotropic support, the mother is critically ill or unable to comply with the follow-up schedule, parental refusal for KMC intervention. Eligible subjects were selected as per inclusion and exclusion criteria. The subjects were divided into two groups; Kangaroo Mother Care (Group-I) and Standard Method Care (Group-II). Randomization was achieved by lottery techniqu
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kangaroo Mother Care (Group-I) (Experimental): In the KMC group mothers were explained detail about KMC adoption in the presence of their family. KMC was initiated as soon as the baby was stable. If the mother is not available initially any of the family members can start KMC. The mother provided skin to skin contact in upright position dressed in a cap, socks, and diaper and supported in the bottom with a sling/binder. Adequate privacy was ensured. Comfortable chairs and beds were provided to the mothers practicing KMC in the nursery. Skin-to-skin contact was given for a minimum of 1 hour at a time and at least for 12 hrs./ day, duration was gradually increased to as long as comfortable to the mother and baby. When the baby is not in KMC, the baby was placed in the cot with adequately clothed and covered. A "KMC" chart was given to the mother to keep a record of the duration of kangaroo care provided. If the mother is unable to fill up the chart, it was done by a close family member.
  Interventions: Other: Kangaroo Mother Care
- Standard Method Care (Group-II) (Active Comparator): Neonate in the SMC group was managed under a radiant warmer.
  Interventions: Other: Standard Medical Care (SMC)

INTERVENTIONS:
Other: Kangaroo Mother Care — Skin-to-skin contact was given for a minimum of 1 hour at a time and at least for 12 hrs./ day, duration was gradually increased to as long as comfortable to the mother and baby.
  Arms: Kangaroo Mother Care (Group-I)
Other: Standard Medical Care (SMC) — In well baby nursery, under radiant warmer
  Arms: Standard Method Care (Group-II)

SUMMARY:
Objective: To compare the outcomes of early kangaroo mother care and standard method care in healthy low birth weight preterm neonates

Introduction:

Globally, prematurity is the leading cause of death in children under the age of 5 years. And in almost all countries with reliable data, preterm birth rates are increasing. Pakistan is leading with prevalence of premature birth as 21.64%. An estimated 15 million babies are born too early every year. That is more than 1 in 10 babies. Approximately 1 million children die each year due to complications of preterm birth. Many survivors face a lifetime of disability, including learning disabilities and visual and hearing problems. The issue of preterm birth is of paramount significance for achieving United Nations Sustainable Development Goal 3 target #3.2, which aims to end all preventable deaths of newborns and children aged under 5 years by 2030.

Preterm low birth weight (LBW) babies are unable to control their body temperature and are at greater risk of illness. Conventional neonatal care of LBW babies is expensive and needs both trained personnel and permanent logistic support like the incubator, warmer etc. Kangaroo Mother Care (KMC) is a special way of caring for low birth weight babies has three main components- (a) thermal care through continuous skin to skin contact (b) support for exclusive breastfeeding (c) early recognition and response to complication. The WHO has defined KMC as early, continuous, and prolonged skin-to-skin contact (SSC) between the mother and preterm babies; exclusive breastfeeding or breast milk feeding; early discharge after hospital-initiated KMC with continuation at home; and adequate support and follow-up for mothers at home. Intermittent KMC was associated with a nearly doubled increase in exclusive breast milk feeding (outcome) and breastfeeding (method) at both discharge and 42 days after discharge for late preterm infants. There is a critical knowledge gap regarding the effect of initiating continuous kangaroo mother care soon after birth and before stabilization with respect to mortality in infants with low birth weight. WHO Immediate KMC study group conducted a large, multicenter, randomized, controlled trial to evaluate the safety and efficacy of continuous kangaroo mother care initiated immediately after birth in infants with a birth weight between 1.0 and 1.799 kg.

Several areas require further study in light of the results of different review studies like methodologically rigorous trials are needed to further explore the effectiveness of early-onset continuous KMC in unstabilized or relatively stabilized LBW infants in low-income settings, to evaluate the use of continuous or intermittent KMC in high-income settings and to report results mainly on infant morbidity, to investigate effects of early-onset KMC on breastfeeding, to assess the cost-effectiveness of KMC in low-, middle-, and high-income settings and to explore the mother-infant attachment. Additional trials in different settings ensuring baseline comparability of mortality, adequate KMC implementation, and birth weight assessment are required to clarify the effect of community-based KMC on LBW neonatal mortality before community-based KMC programs are implemented and before community-based KMC is included in essential newborn care.

This study is conducted to compare the outcomes in healthy low birth weight preterm infants managed through early kangaroo mother care in first 24 hours of birth and standard methods of care.

Inclusion criteria:

Inclusion criteria are as follows:

New admission of singleton or twin (inborn or out-born) Weight < 2000 g (as per study scale) Age 1-24 h old when screening begins Gestational age >30 weeks to <37 weeks Mother or other caregiver available and willing to provide intervention

Exclusion criteria:

Exclusion criteria are as follows:

Triplets who are all admitted to the study site Congenital malformation not compatible with life or needing immediate surgical intervention Severe jaundice Seizures Stable as assessed during cardio-respiratory screening Severely unstable as assessed during cardio-respiratory screening or died during screening Severe perinatal asphyxia Babies require a ventilator or inotropic support The mother is critically ill or unable to comply with the follow-up schedule No study bed available Neonates/mothers enrolled in another research study No written informed consent from parent or caregiver within 24 h of admission. Study type: Randomized controlled trial Study population: Low birth weight healthy preterm infants born at gynecology department of Services Hospital Lahore

ELIGIBILITY:
Inclusion Criteria:

* New admission of singleton or twin (inborn or out-born)
* Weight < 2000 g (as per study scale)
* Age 1-24 h old when screening begins
* Gestational age >30 weeks to <37 weeks
* Mother or other caregiver available and willing to provide intervention

Exclusion Criteria:

* Triplets who are all admitted to the study site
* Congenital malformation not compatible with life or needing immediate surgical intervention
* Severe jaundice
* Seizures
* Stable as assessed during cardio-respiratory screening
* Severely unstable as assessed during cardio-respiratory screening or died during screening
* Severe perinatal asphyxia
* Babies require a ventilator or inotropic support
* The mother is critically ill or unable to comply with the follow-up schedule
* No study bed available
* Neonates/mothers enrolled in another research study
* No written informed consent from parent or caregiver within 24 h of admission.

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Number of neonatal deaths within 72 hours after enrollment | 0-72 hours of age
  Vital status will be assessed every 12 hours during hospital stay. Neonatal death is defined as cessation of breathing and circulation confirmed by attending physician.
Number of neonatal deaths within 28 days of age | Enrollment to Day 28
  Vital status assessed every 12 hours during hospitalization and via home visit on Day 29.
Length of hospital stay from enrollment to discharge | Enrollment to discharge
  Total days spent in nursery/KMC ward from admission to discharge as documented in hospital records.

SECONDARY OUTCOMES:
Number of infants exclusively breastfed at 29 days of age | Day 29
  Assessed via 24-hour feeding recall during home visit. Exclusive breastfeeding means no other liquids or solids except prescribed medicines/supplements.
Number of infants with clinically suspected sepsis during hospital stay | Enrollment to discharge/Day 28
  Suspected sepsis identified through 12-hourly clinical records and laboratory evaluation based on unit protocol.

OTHER OUTCOMES:
Maternal satisfaction score with hospital care | At discharge
  Structured interview-based rating of overall hospital care experience by the mother.
Maternal depressive symptoms using PHQ-9 scale | Day 29
  Mother scores ≥15 considered depressed as per PHQ-9 validated cutoff.

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital and Medical Centre, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Due to confidentiality